CLINICAL TRIAL: NCT02996448
Title: A Phase 2a Study to Evaluate the Safety, Tolerability, and Immunogenicity of One Dose of NDV-3A Vaccine in Patients With STAT3-Mutated Hyper-IgE Syndrome
Brief Title: Safety, Tolerability, and Immunogenicity of One Dose of NDV 3A Vaccine in People With STAT3-Mutated Hyper-IgE Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety concerns led to early termination.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 170017; 17-I-0017
Record Dates: First submitted 2016-12-16; First posted 2016-12-19 (Estimated); Results first posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2018-10

CONDITIONS: Autosomal-dominant Hyper-IgE Syndrome
Keywords: AD-HIES; Anti-rAls3 Antibody; Staphylococcus Aureus; Candida Albicans; RNA Transcriptome
MeSH Terms: conditions — Job Syndrome; Staphylococcal Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (1):
- NDV 3A vaccine (Experimental): Participants will receive a single dose of 0.5 mL (300 micrograms of rAls3) administered via IM injection.
  Interventions: Drug: NDV-3A

INTERVENTIONS:
Drug: NDV-3A — A vaccine containing recombinant Candida albicans agglutinin-like sequence 3 (rAls3) protein as the antigen, formulated with AlOH adjuvant in phosphate buffered saline. Participants will receive a single 0.5 mL dose containing 300 micrograms of rAls3 and 0.5 mg of aluminum as AlOH, delivered via intramuscular injection.

SUMMARY:
Background:

AD-HIES is a disease that weakens the immune system. It puts people at risk for infections, particularly Staph and Candida infections. Researchers want to test a vaccine that may help keep people from getting these infections, which would help people with AD-HIES.

Objective:

To test the new vaccine NDV-3A for protection against infection from the yeast Candida and the bacterium Staphylococcus aureus (Staph).

Eligibility:

Adults ages 18-55 who have AD-HIES

Healthy volunteers ages 18-55

Design:

Participants will have 6-7 study visits over 6-7 months. They will also be contacted by phone in between some visits.

Participants will be screened with a medical history, physical exam, and blood and urine tests.

Participants will have 2 baseline visits. They will have repeat the screening tests. They will have samples of saliva, stool, skin, mucus (oral, nasal, and/or vaginal) collected. Vaginal and stool samples are optional. Any eczema on their skin will be looked at.

Participants will fill out symptom diary cards to record how they feel.

Participants will have the NDV-3A vaccine injected into a muscle in the arm.

Participants will return the next 2 days. They will have a physical exam. Blood will be collected.

Participants will have 2 more follow-up visits at the NIH. They will have a physical exam. They will have blood, saliva, stool, skin, vaginal fluid, and/or mucus samples collected. Vaginal and stool samples are optional.

Participants will be called once a month for 5 months after the vaccination. There is an optional visit about 6 weeks after the vaccination. Participants will provide a blood sample at this visit.

DETAILED DESCRIPTION:
Autosomal-dominant hyper-IgE syndrome (AD-HIES) is characterized by recurrent Staphylococcus aureus and Candida epithelial infections, which is thought to be due, in part, to a lack of Th17 cell differentiation, thus impairing epithelial immunity. Treatment of AD-HIES is primarily supportive with prophylactic antibiotics; however, this is limited by microbial resistance and intolerance of medications, and infections do still occur. Immunological intervention with a vaccine could improve quality of life by preventing these infections altogether.

The NDV-3A vaccine consists of a recombinant protein derived from the Candida Als3 adhesion protein. This protein is homologous to surface proteins on S aureus and has been shown in preclinical studies to protect against both intravascular and subcutaneous challenge with S aureus. Therefore, NDV-3A represents not only the first antifungal vaccine, but also the first vaccine to provide cross-kingdom protection. In Phase 1 and Phase 2 studies in healthy volunteers (150 receiving vaccine), the safety profile of this vaccine is very reassuring as the vaccine elicits a strong antibody response after a single dose in all vaccinees as well as a Th1 and/or Th17 response in the majority of vaccinees. We will enroll 20 healthy adult volunteers and 20 adults with AD-HIES in an open-label, single-dose study to assess the immunological response to and the safety/tolerability of the NDV-3A vaccine. We anticipate an increase in baseline anti-Als3 IgG within 2 weeks post-vaccination.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age 18-55 years.
  2. For healthy volunteers: in general good health, without significant medical illness, physical exam findings, or significant laboratory abnormalities as determined by the investigator.
  3. For participants with AD-HIES: confirmation of diagnosis with a STAT3 mutation.
  4. Participants who can get pregnant must be willing to use an acceptable form of contraception for the duration of participation and have a negative pregnancy test at screening.
  5. Agree to allow storage of biological samples for future research.

EXCLUSION CRITERIA:

1. Has a history of allergic response or other serious reaction to aluminum and/or yeast products.
2. Has a history of clinically significant allergy including anaphylaxis or other serious reaction to food, vaccines, or other drugs, that in the opinion of the investigator, might put the participant at undue risk.
3. Has an active infection (such as S aureus abscess, pneumonia, acute Candida mucocutaneous infection). Baseline state of chronic infections will be considered by the PI (eg, chronic Pseudomonas infection in lung).
4. Has an active infection with hepatitis B, hepatitis C, or HIV.
5. Has received or is planning to receive any investigational drug, investigational vaccine, or investigational device within four weeks prior to vaccination, or at any other time during their participation in the study.
6. Has received or is planning to receive any other live vaccine within three weeks before vaccination or for three weeks after vaccination.
7. Self-reported current alcohol abuse or addiction.
8. Self-reported current illicit drug abuse or addiction, or drug screen positive for illicit drugs.
9. Current or planned use, within 3 weeks before vaccination, of any medications or treatments that may alter immune responses to the study vaccine (eg, immunosuppressive medications including systemic corticosteroids, cyclosporine, tacrolimus, cytotoxic drugs, Bacillus Calmette-Guerin, monoclonal antibodies, or radiation therapy). Topical, intranasal, or inhaled immunosuppressants such as corticosteroids will be allowed.
10. Current or planned use within 2 weeks before vaccination of immune globulin replacement.
11. Has any of the following laboratory abnormalities at the screening visit:

    1. Alanine transaminase (ALT), aspartate transaminase (AST), and/or alkaline

       phosphatase (ALP) > 1.5 times the upper limit of normal (ULN).
    2. Total bilirubin level > 1.5 times the ULN
    3. Serum creatinine level > 1.5 times the ULN
    4. Absolute neutrophil count < 750 cells/microliter
    5. Hemoglobin < 9 mg/dL
    6. Platelet count < 100,000
12. Refusal or inability to comply with study procedures to the extent that it is potentially harmful to the participant or to the integrity of the study data.
13. Has donated blood/plasma within four weeks before vaccination.
14. Is pregnant or breastfeeding, or intends to become pregnant over the course of the study.
15. Is unable to commit to the follow-up visits and or has unreliable access to a telephone for follow-up contacts, either by self-admission (self-reporting) or in the opinion of the investigator.
16. Any other condition the investigator believes would interfere with the participant s ability to provide informed consent, comply with study instructions, or that might confound the interpretation of the study results or put the participant at undue risk.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2016-11-17; Primary Completion 2018-07-22 (Actual); Study Completion 2018-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Freeman, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sowerwine KJ, Holland SM, Freeman AF. Hyper-IgE syndrome update. Ann N Y Acad Sci. 2012 Feb;1250:25-32. doi: 10.1111/j.1749-6632.2011.06387.x. Epub 2012 Jan 23. PMID 22268731
- [Background] Spellberg BJ, Ibrahim AS, Avanesian V, Fu Y, Myers C, Phan QT, Filler SG, Yeaman MR, Edwards JE Jr. Efficacy of the anti-Candida rAls3p-N or rAls1p-N vaccines against disseminated and mucosal candidiasis. J Infect Dis. 2006 Jul 15;194(2):256-60. doi: 10.1086/504691. Epub 2006 Jun 6. PMID 16779733
- [Background] Liu Y, Filler SG. Candida albicans Als3, a multifunctional adhesin and invasin. Eukaryot Cell. 2011 Feb;10(2):168-73. doi: 10.1128/EC.00279-10. Epub 2010 Nov 29. PMID 21115738
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-I-0017.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Healthy volunteers were not enrolled to the study due to the early termination. The three subjects enrolled were those with AD-HIES.
Groups:
- Vaccination Group, Single Arm Study: Participants will receive a single dose of 0.5 mL (300 micrograms of rAls3) administered via IM injection.
  NDV-3A: A vaccine containing recombinant Candida albicans agglutinin-like sequence 3 (rAls3) protein as the antigen, formulated with AlOH adjuvant in phosphate buffered saline. Participants will receive a single 0.5 mL dose containing 300 micrograms of rAls3 and 0.5 mg of aluminum as AlOH, delivered via intramuscular injection.
Period: Overall Study
Arm/Group | Vaccination Group, Single Arm Study
Started | 3
Completed | 0
Not Completed | 3
Not completed — Study terminated due to adverse effects | 3

BASELINE CHARACTERISTICS:
Groups:
- Vaccination Group- Single Arm Study: Participants will receive a single dose of 0.5 mL (300 micrograms of rAls3) administered via IM injection.
  NDV-3A: A vaccine containing recombinant Candida albicans agglutinin-like sequence 3 (rAls3) protein as the antigen, formulated with AlOH adjuvant in phosphate buffered saline. Participants will receive a single 0.5 mL dose containing 300 micrograms of rAls3 and 0.5 mg of aluminum as AlOH, delivered via intramuscular injection.
Arm/Group | Vaccination Group- Single Arm Study
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 20 [19 to 26]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent of Each Group With at Least a Four-fold Increase in Anti rAls3 Antibody Titer.
Description: Antibody titer
Time Frame: 2 weeks after vaccination
Population: As study was stopped prematurely due to safety concerns, the data was not obtained.
Groups:
- Vaccine Recipients: Participants will receive a single dose of 0.5 mL (300 micrograms of rAls3) administered via IM injection.
  NDV-3A: A vaccine containing recombinant Candida albicans agglutinin-like sequence 3 (rAls3) protein as the antigen, formulated with AlOH adjuvant in phosphate buffered saline. Participants will receive a single 0.5 mL dose containing 300 micrograms of rAls3 and 0.5 mg of aluminum as AlOH, delivered via intramuscular injection.
Arm/Group | Vaccine Recipients
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Serious Adverse Events That Led to Study Termination.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccination Group- Single Arm Study
Number analyzed (Participants) | 3
Participants | 1

3. Secondary Outcome: Anti-Als3 Antibody Titers at 6 Months After Vaccination in Patients With AD HIES and Healthy Volunteers.
Time Frame: 6 months
Population: Data were not collected due to premature termination of study.
Arm/Group | Vaccination Group- Single Arm Study
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Vaccination Group- Single Arm Study
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccination Group- Single Arm Study (N=3)
Anaphylaxis (Immune system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccination Group- Single Arm Study (N=3)
Injection site pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Dizziness (Nervous system disorders) | 1
fatigue (Nervous system disorders) | 1
Eczema exacerbation (Skin and subcutaneous tissue disorders) | 2
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/48/NCT02996448/Prot_SAP_000.pdf